CLINICAL TRIAL: NCT01613378
Title: A Multi-National, Multi-Center Non-Interventional Study in Rheumatoid Arthritis (RA) Patients Who Are Treated With Tocilizumab
Brief Title: A Non-Interventional Study in Rheumatoid Arthritis Patients Treated With Tocilizumab (RoActemra/Actemra)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28121
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Results first posted 2016-10-04 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Rheumatoid Arthritis Cohort: The cohort included participants with moderate to severe rheumatoid arthritis (RA) in whom the treating physician made the decision to initiate tocilizumab treatment.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention administered in this study

SUMMARY:
This multi-center, non-interventional study will evaluate the pattern of usage in clinical practice, efficacy and safety of tocilizumab in patients with rheumatoid arthritis. Patients initiated on treatment with tocilizumab according to the licensed Canadian product monograph recommendations will be followed for 12 months from the start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Moderate to severe rheumatoid arthritis according to revised (1987) American college of rheumatology (ACR) criteria
* Initiated on tocilizumab treatment by the treating physician in accordance with the Canadian product monograph
* Informed consent to data being subject to computerized data processing
* Participant must fulfill the reimbursement criteria for treatment with tocilizumab under provincial or private health insurance coverage

Exclusion Criteria:

* Received tocilizumab prior to enrolment visit
* Previously received tocilizumab in a clinical trial or for compassionate use
* Enrolled in an ongoing clinical trial and/or received treatment with any investigational agent within 4 weeks, or 5 half-lives of the investigational agent, whichever is longer, before starting treatment with tocilizumab
* Participation in another clinical trial or industry sponsored observational study
* History of autoimmune disease or any joint inflammatory disease other than rheumatoid arthritis, with the exception of concomitant secondary Sjörgen's syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population included participants with moderate to severe rheumatoid arthritis (RA) in whom the treating physician made the decision to initiate tocilizumab treatment.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (27):
- Canada (27):
  - Edmonton, Alberta
  - Kelowna, British Columbia
  - Nanaimo, British Columbia
  - Penticton, British Columbia
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - St. John's, Newfoundland and Labrador
  - Lunenburg, Nova Scotia
  - Sydney, Nova Scotia
  - Brampton, Ontario
  - Burlington, Ontario
  - Hamilton, Ontario
  - Markham, Ontario
  - Mississauga, Ontario
  - Newmarket, Ontario
  - St. Catharines, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
  - Laval, Quebec
  - Montreal, Quebec
  - Pointe-Claire, Quebec
  - Québec, Quebec
  - Rimouski, Quebec
  - Saint-Eustache, Quebec
  - Sherbrooke, Quebec
  - Trois-Rivières, Quebec
  - Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Haraoui B, Jamal S, Ahluwalia V, Fung D, Manchanda T, Khraishi M. Real-World Tocilizumab Use in Patients with Rheumatoid Arthritis in Canada: 12-Month Results From an Observational, Noninterventional Study. Rheumatol Ther. 2018 Dec;5(2):551-565. doi: 10.1007/s40744-018-0130-6. Epub 2018 Oct 28. PMID 30370468

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rheumatoid Arthritis Cohort
Started | 200
Completed | 161
Not Completed | 39
Not completed — Lack of Efficacy | 13
Not completed — Adverse Event | 11
Not completed — Withdrawal by Subject | 8
Not completed — Death | 2
Not completed — Lost to Follow-up | 1
Not completed — Other Reason | 4

BASELINE CHARACTERISTICS:
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.43 (13.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants on Tocilizumab Treatment at 6 Months After Treatment Initiation
Time Frame: At 6 months
Population: All participants enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 200
percentage of participants | 81.5 [75.4 to 86.6]

2. Secondary Outcome: Change From Baseline in Tender Joint Count (TJC)
Description: Following an assessment of 68 joints for tenderness, joints were classified as tender or not tender by the investigator.
Time Frame: From baseline to Month 12
Population: Full analysis set (FAS) population consisted of all participants included in the study who received at least one dose of Tocilizumab (n=198). Only participants who completed the Tender Joint Count were included in this analysis.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 146
tender joints | -12.71 (12.84)

3. Secondary Outcome: Change From Baseline in Swollen Joint Count (SJC)
Description: Following an assessment of 66 joints for swelling, joints were classified as swollen or not swollen by the investigator.
Time Frame: From baseline to Month 12
Population: Full analysis set (FAS) population consisted of all participants included in the study who received at least one dose of Tocilizumab (n=198). Only participants who completed the Swollen Joint Count were included in this analysis.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 146
swollen joints | -8.66 (7.67)

4. Secondary Outcome: Change From Baseline in Disease Activity Score 28 (DAS28)
Description: The DAS28 scale is a combined index for measuring disease activity in rheumatoid arthritis. Scores range from 0 to 10, with higher scores representing more disease activity.
Time Frame: From baseline to Month 12
Population: Full analysis set (FAS) population consisted of all participants included in the study who received at least one dose of Tocilizumab (n=198). Only participants who completed the DAS28 assessment were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 117
units on a scale | -3.00 (1.73)

5. Secondary Outcome: Change From Baseline in Duration of Morning Stiffness (Visual Analog Scale, VAS)
Description: With VAS, participants specify their level of agreement to a statement by indicating a position along a continuous line between two endpoints, with 0 being the lowest level and 100 being the highest level of morning stiffness.
Time Frame: From baseline to Month 12
Population: Full analysis set (FAS) population consisted of all participants included in the study who received at least one dose of Tocilizumab (n=198). Only participants who completed the assessment of Duration of Morning Stiffness on the VAS were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 143
units on a scale | -24.31 (30.04)

6. Secondary Outcome: Change From Baseline in Patient Global Assessment of Disease Activity (Visual Analog Scale, VAS)
Description: With VAS, participants specify their level of agreement to a statement by indicating a position along a continuous line between two endpoints, with 0 being the lowest level and 100 being the highest level of disease activity.
Time Frame: From baseline to Month 12
Population: Full analysis set (FAS) population consisted of all participants included in the study who received at least one dose of Tocilizumab (n=198). Only participants who completed the Assessment of Disease Activity on the VAS were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 144
units on a scale | -24.90 (29.30)

7. Secondary Outcome: Change From Baseline in Physician Global Assessment of Disease Activity (Visual Analog Scale, VAS)
Description: With VAS, physicians specify their level of agreement to a statement by indicating a position along a continuous line between two endpoints, with 0 being the lowest level and 100 being the highest level of disease activity.
Time Frame: From baseline to Month 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 157
units on a scale | -39.95 (28.28)

8. Secondary Outcome: Change From Baseline in Patient Assessment of Pain (Visual Analog Scale, VAS)
Description: With VAS, participants specify their level of agreement to a statement by indicating a position along a continuous line between two endpoints, with 0 being the lowest level and 100 being the highest level of pain.
Time Frame: From baseline to Month 12
Population: Full analysis set (FAS) population consisted of all participants included in the study who received at least one dose of Tocilizumab (n=198). Only participants who completed the Assessment of Pain on the VAS were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 144
units on a scale | -27.99 (30.47)

9. Secondary Outcome: Change From Baseline in Patient Assessment of Fatigue (Visual Analog Scale, VAS)
Description: With VAS, participants specify their level of agreement to a statement by indicating a position along a continuous line between two endpoints, with 0 being the lowest level and 100 being the highest level of fatigue.
Time Frame: From baseline to Month 12
Population: Full analysis set (FAS) population consisted of all participants included in the study who received at least one dose of Tocilizumab (n=198). Only participants who completed the Patient Assessment of Fatigue on the VAS were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 143
units on a scale | -23.94 (30.55)

10. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP)
Description: The serum concentration of C-reactive protein (CRP) was measured. A reduction in the level of CRP was considered an improvement.
Time Frame: From baseline to Month 12
Population: Full analysis set (FAS) population consisted of all participants included in the study who received at least one dose of Tocilizumab (n=198). Only participants who completed the CRP assessment were included in this analysis.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 120
mg/L | -16.35 (31.68)

11. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR)
Description: The erythrocyte sedimentation rate (ESR) was analyzed at the site using the kit provided by the central laboratory. A reduction in the level of ESR was considered an improvement.
Time Frame: From baseline to Month 12
Population: Full analysis set (FAS) population consisted of all participants included in the study who received at least one dose of Tocilizumab (n=198). Only participants who completed the ESR assessment were included in this analysis.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 104
mm/hr | -16.79 (22.71)

12. Secondary Outcome: Percentage of Participants With Changes in Extra-Articular Manifestations at 12 Months
Description: The extra-articular RA manifestations ascertained were the nodules, Raynaud's phenomenon, secondary Sjogren's syndrome, pulmonary fibrosis, pericarditis, polyneuropathy, scleritis, severe cutaneous vasculitis, weight loss and anemia. Percentages are based on the total number of participants with available data.
Time Frame: At 12 months
Population: Full analysis set (FAS) population consisted of all participants included in the study who received at least one dose of Tocilizumab (n=198). Only participants who completed the assessment of Extra-Articular Manifestations were included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 161
percentage of participants
  Nodules | 3.1
  Raynaud"s Phenomenon | 0
  Secondary Sjogren"s Syndrome | 2.5
  Pulmonary Fibrosis | 0
  Pericarditis | 0
  Polyneuropathy | 0
  Scleritis | 0
  Severe Cutaneous Vasculitis | 0
  Weight Loss | 0.6
  Anemia | 1.2

13. Secondary Outcome: Number of Participants With Changes in Severity of Extra-Articular Manifestations at 12 Months
Description: The severity of extra-articular RA manifestations ascertained were the nodules, Raynaud's phenomenon, secondary Sjogren's syndrome, pulmonary fibrosis, pericarditis, polyneuropathy, scleritis, severe cutaneous vasculitis, weight loss and anemia. Percentages are based on the total number of participants who responded "YES" to changes in extra- articular RA manifestations (new presence or change in severity) since the last visit. NA=Not applicable
Time Frame: At 12 months
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 161
participants
  Nodules: Mild | 5
  Nodules: Moderate | 0
  Nodules: Severe | 0
  Raynaud"s Phenomenon: Mild | NA — No change was evident.
  Secondary Sjogren"s Syndrome: Mild | 3
  Secondary Sjogren"s Syndrome: Moderate | 1
  Secondary Sjogren"s Syndrome: Severe | 0
  Pulmonary Fibrosis: Moderate | NA — No change was evident.
  Pulmonary Fibrosis: Severe | NA — No change was evident.
  Pericarditis: Mild | NA — No change was evident.
  Severe Cutaneous Vasculitis: Mild | NA — No change was evident.
  Severe Cutaneous Vasculitis: Moderate | NA — No change was evident.
  Weight Loss: Mild | 1
  Weight Loss: Moderate | 0
  Weight Loss: Severe | 0
  Anemia: Mild | 2
  Anemia: Moderate | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Rheumatoid Arthritis Cohort
Serious Adverse Events (participants affected / at risk) | 31/198
Other Adverse Events (participants affected / at risk) | 68/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rheumatoid Arthritis Cohort (N=198)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Chest discomfort (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Mass (General disorders) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Postoperative wound infection (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Hypersensitivity vasculitis (Vascular disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Fat embolism (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint instability (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Bladder prolapse (Renal and urinary disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1)
Obstructive shock (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rheumatoid Arthritis Cohort (N=198)
Nausea (Gastrointestinal disorders) | 10 (11)
Fatigue (General disorders) | 10 (11)
Bronchitis (Infections and infestations) | 10 (10)
Upper respiratory tract infection (Infections and infestations) | 23 (30)
Urinary tract infection (Infections and infestations) | 10 (17)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 10 (13)
Headache (Nervous system disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.